CLINICAL TRIAL: NCT06678711
Title: Randomized Controlled Study of Minimally Invasive Atlantoaxial Mass Fusion and Open Atlantoaxial Fusion in the Treatment of Atlantoaxial Dislocation
Brief Title: Minimally Invasive Atlantoaxial Lateral Mass Joint Fusion (MIS-PALF) As a Surgical Treatment of Atlantoaxial Dislocation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Hebei Medical University Third Hospital (Other); Shanxi Bethune Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Tianjin People's Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Daping Hospital of Army Medical University (Other); Shengjing Hospital (Other); The Third Bethune Hospital of Jilin University (Unknown)
Responsible Party: Principal Investigator, Wang Shenglin, Clinical Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2024730
Record Dates: First submitted 2024-11-02; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Atlantoaxial Dislocation
Keywords: atlantoaxial dislocation; MIS-PALF; minimal invasive surgery
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimal invasive surgery arm (Experimental): Patients in minimal invasive surgery arm will receive minimal invasive surgery-posterior atlantoaxial lateral mass joint fusion.
  Interventions: Procedure: minimal invasive surgery-posterior atlantoaxial lateral mass joint fusion
- Open atlantoaxial fixation and fusion arm (Active Comparator): Patients in open atlantoaxial fixation and fusion arm will receive atlantoaxial fixation and fusion using the Goel-Harms technique.
  Interventions: Procedure: Open atlantoaxial fixation and fusion

INTERVENTIONS:
Procedure: minimal invasive surgery-posterior atlantoaxial lateral mass joint fusion — Make a 4.5 cm incision along the median line and then dissect the trapezius, splenius capitis, and semispinalis capitis muscle laterally 1.5 cm off the median line. Retract the obliquus capitis inferior muscle to expose the C1-C2 intra-articular space. Remove the articular cartilage, insert allogenic granular bone and 3D-printed cage. Place the screws and rod in the same positions as conventional surgery, and the operation is completed.
  Arms: Minimal invasive surgery arm
Procedure: Open atlantoaxial fixation and fusion — The Goel-Harms procedure will be used in the control group. Screws and rods are placed in the same position as in the experimental group, and a negative-pressure drain was placed until daily drainage was <50 mL.
  Arms: Open atlantoaxial fixation and fusion arm

SUMMARY:
The conventional treatment for atlantoaxial dislocation is atlantoaxial fixation and fusion using the Goel-Harms technique, which involves a midline incision, dissection of the occipital muscle group, and is associated with disadvantages such as damage to the posterior ligament and muscle, high incidence of postoperative occipital cervical pain, and significant blood loss due to intraoperative bleeding and postoperative drainage. Since 2013, various studies have reported minimally invasive posterior atlantoaxial lateral mass joint fusion techniques through muscle spaces, but previous studies were all case reports, without sufficient reliability and controlled studies. The Department of Orthopedics at Peking University Third Hospital has been using the minimal invasive surgery-posterior atlantoaxial lateral mass joint fusion (Mis-PALF) technique for the treatment of atlantoaxial dislocation since 2015, with preliminary good clinical results. In order to further compare the advantages and disadvantages of the two surgical methods from a larger sample, a randomized controlled study is planned. The patients will be randomly divided into two groups, with the experimental group receiving the Mis-PALF surgery and the control group receiving open atlantoaxial fusion and fixation. There will be a 1-2 year follow-up to compare the safety and effectiveness of the two surgical methods for the treatment of atlantoaxial dislocation.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 0 to 80 years old, regardless of gender
2. Diagnosed with atlantoaxial dislocation, suitable for posterior surgical treatment
3. Index of assessment integrity
4. Agree to participate in the study and sign the informed consent

Exclusion Criteria:

1. Atlantoaxial dislocation without surgical treatment
2. Atlantoaxial dislocation treated by other operation, such as TARP

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative Blood Loss | 2 weeks
  Blood loss due to intraoperative bleeding and postoperative drainage.
Postoperative Stay | 2 weeks
  The time from the completion of surgery to the patient leaving hospital.
Level of Occipitocervical Pain | 12 months
  The level of patients' occipitocervical pain is described by Numerical Rating Scale, from zero to ten, and ten means the most pain.
Main location of occipitocervical pain | 12 months
  The location of patients' occipitocervical pain is indicated by patients on a diagram illustrating the anatomical regions of the head and neck.
Painkillers Used for Occipitocervical Pain | 12 months
  Patients are asked about whether they used any painkillers for occipitocervical pain and which painkillers they used.

SECONDARY OUTCOMES:
Incidence of Adverse Events | 12 months
  This metric is defined as the proportion of adverse events that manifest during the study's duration relative to the total number of patients enrolled. Adverse events encompass a range of critical factors, including but not limited to: Neurological deterioration, Incision infection, Vascular injury, Airway obstruction, Poor reduction, Unplanned readmission and re-surgery, Internal fixation failure, Fusion failure, Surgical-related lower cervical spine deformities.
Atlantoaxial Reduction Rate | 12 months
  To gauge the effectiveness of the surgical interventions in achieving atlantoaxial reduction, postoperative CT scans of the head and neck will be conducted. Measurements will be taken of the distance between the odontoid process and key reference lines, including Chamberlain's line (CL), Wackenheim line (WL), McRae line (ML), and atlantodental interval (ADI). The reduction rate will be calculated by comparing the postoperative measurements to the preoperative values, expressed as a ratio.
Bone Graft Fusion Rate | 12 months
  Evaluation of the proportion of patients exhibiting successful bone fusion between the atlas and axis will be conducted through postoperative three-dimensional CT examinations of the cervical spine. The bone graft fusion rate will be determined by calculating the number of patients with evident fusion relative to the total number of patients enrolled.
Improvement Rate of Quality of Life | 12 months
  The quality of life for each patient will be assessed using the Short Form 12-Item(SF-12) Health Survey. SF-12 scores ranges from 0 to 100, and 100 usually means healthier in a certain dimension. The improvement rate in quality of life will be calculated based on the preoperative and postoperative differences in SF-12 scores. This indicator offers insights into the impact of surgical interventions on patients' overall well-being and quality of life, providing a vital perspective on treatment effectiveness.
Improvement of Neurological Function | 12 months
  To assess the extent of neurological function improvement, patients' Japanese Orthopaedic Association(JOA) scores one year after surgery will be compared with their preoperative scores. JOA score ranges form 0 to 17, and 0 means worse neurological function. The JOA improvement rate will be calculated based on the cervical JOA score, employing the Hirabayashi method formula: JOA Improvement Rate = (Postoperative JOA Score - Preoperative JOA Score) / (17 - Preoperative JOA Score) * 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No